CLINICAL TRIAL: NCT00006402
Title: Lifestyle, Adiposity and Cardiovascular Health in Youths
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 927
Record Dates: First submitted 2000-10-12; First posted 2000-10-13 (Estimated); Last update posted 2008-01-21 (Estimated); Status verified 2008-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity

SUMMARY:
To determine the influences of diet and physical activity (PA) on total body fatness and regional fat distribution and the relationship of these to risk factors of cardiovascular disease during adolescence.

DETAILED DESCRIPTION:
BACKGROUND:

Adult studies have shown that adiposity, especially visceral adipose tissue, and cardiovascular (CV) fitness are key links between lifestyle factors like diet and exercise on one hand, and CV disease on the other. However, very little is known about these links during the juvenile years, when the processes leading to CV disease are at an early stage of development.

The study is in response to a Program Announcement issued in March 1998 on Diet and Cardiovascular Disease Risk in Children and Adolescents. The Program Announcement, jointly issued by the National Institute of Nursing Research and the NHLBI, sought to encourage research relevant to the development and/or testing of dietary interventions to improve the cardiovascular disease (CVD) risk profiles in children and adolescents, especially those at increased risk for CVD or for development of CVD risk factors because of genetics, family history, socioeconomic status (SES), race/ethnicity, levels of blood cholesterol or blood pressure, or other factors.

DESIGN NARRATIVE:

The study determines the relations of free-living diet and exercise to total body percent fat ( percent BF), visceral adipose tissue and CV fitness in black and white boys and girls of varying socioeconomic status (SES). The study also determines the relations of fatness and fitness to different CVD risk factors. A total of 800 15 to 18 year olds, 200 in each ethnic and gender subgroup will be recruited. Diet will be assessed with seven 24-hour recalls, and exercise with two seven-day recalls and heart rate monitoring. Percent body fat will be measured with dual-energy x-ray absorptiometry, visceral adipose tissue with magnetic resonance imaging and CV fitness with a multi-stage treadmill test. Measurements will be made of major fatness- and fitness-related CV disease risk factors (e.g., total cholesterol:HDL cholesterol ratio, insulin, systolic blood pressure, left ventricular mass indexed to height, fibrinogen). Multivariate and univariate analyses will be conducted to determine relationships.

ELIGIBILITY:
No eligibility criteria

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2000-08; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paule Barbeau — Augusta University

REFERENCES:
- [Background] Litaker MS, Barbeau P, Humphries MC, Gutin B. Comparison of Hologic QDR-1000/W and 4500W DXA Scanners in 13- to 18-Year Olds. Obes Res. 2003 Dec;11(12):1545-52. doi: 10.1038/oby.2003.206. PMID 14694220